CLINICAL TRIAL: NCT05485701
Title: Perinatal Mental Health Study (PMHS): a Cohort and Validation Study in Two Low-income Settings in India
Brief Title: Perinatal Mental Health Study (PMHS) India
Acronym: PMHS
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: National Institute of Mental Health and Neuro Sciences, India (Other); Dr. Rajendra Prasad Government Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: 10-20
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Depression; Anxiety; Suicidal Ideation; Somatization; PTSD
Keywords: Perinatal; Post-partum; Antenatal; Low- and middle-income country; India; Common mental disorders; Screening; Validation; Prevalence; Risk factor
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicidal Ideation; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perinatal women: Women will be recruited in their first trimester of pregnancy and followed-up until 6 months post-partum. This is the 'exposed' group.
  Interventions: Diagnostic Test: Screening tools for common mental disorders
- Non-perinatal women: Non-perinatal women will be recruited as the 'non-exposed' group and followed-up over the same duration as the perinatal group.
  Interventions: Diagnostic Test: Screening tools for common mental disorders

INTERVENTIONS:
Diagnostic Test: Screening tools for common mental disorders — A number of screening tools will be administered which will establish the likelihood of depression, anxiety, PTSD, somatisation and suicidality.

SUMMARY:
The purpose of this observational study is to improve understanding of mental disorders among perinatal women in India.

DETAILED DESCRIPTION:
The purpose of this observational study is to assess the mental health of perinatal women living in two low-income settings in India. The first phase will explore women's awareness of mental illness and acceptability of screening for mental disorders. The second phase will be a validation study, during which the psychometric properties of screening tools will be assessed against a gold standard. The third stage will comprise a cohort study, during which the prevalence of and risk factors for mental disorders among perinatal and non-perinatal women will be established.

ELIGIBILITY:
Inclusion Criteria:

For Phase 1 (qualitative study) and Phase 2 (validation study):

Pregnant women:

* Aged 18 to 45 years
* Currently pregnant (any trimester)
* Willing and able to give informed consent

Post-partum women:

* Aged 18 to 45 years
* Currently post-partum (between 1-12 months postpartum)
* Willing and able to give informed consent

Non-perinatal women:

* Aged 18 to 45 years
* Not currently pregnant and not given birth in the past 12 months
* Willing and able to give informed consent

For Phase 3 (prospective cohort study):

Perinatal women:

* Aged 18 to 45 years
* In early pregnancy (estimated gestational age <20 weeks) at recruitment
* Not planning to relocate for the duration of the study period
* Willing and able to give informed consent
* Expressed a willingness to continue to participate for the four planned visits

Non-perinatal women:

* Aged 18 to 45 years
* Not currently pregnant and not given birth in the last 12 months
* Not planning to relocate for the duration of the study period
* Willing and able to give informed consent
* Expressed a willingness to continue to participate for the four planned visits

Exclusion Criteria:

The participant may not enter the study if:

* They have an acutely severe psychiatric illness which impairs their ability to take part in the study
* They are not willing or able to provide informed consent

Other than for current severe psychiatric illness which affects ability to participate in the study, we will not exclude any participant on the basis of current or prior physical, psychological or psychiatric co-morbidities so long as she is willing to participate, her ability to take part is not compromised and her ability to give informed consent is not impaired by these conditions.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study participants are women aged 18-45 years living in two low-income settings who fall into one of the following groups:
  (i) pregnant women: women who are pregnant (any trimester of pregnancy) (ii) post-partum women: women who are within 12 months post-partum (iii) non-perinatal women: women who are not currently pregnant and have not given birth within the past 12 months
Sampling Method: Non-Probability Sample
Enrollment: 2332 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Codes and themes relating to acceptability of screening for perinatal mental disorders | To be completed by August 2022
  These will be themes emerging from focus groups with women around awareness of perinatal mental disorders and acceptability of screening.
Phase 2: Psychometric properties of screening tools for common mental disorders | September 2022 - August 2023
  The psychometric properties (sensitivity, specificity, area under the receiver operating curve, optimal cut-off and accuracy) of eight screening tools in Kannada and Hindi will be established among three groups of women: pregnant, post-partum and non-perinatal.
Phase 3: Point prevalence, period prevalence and incidence (with 95% confidence intervals) of common mental disorders among perinatal and non-perinatal women | September 2023 - August 2024
  During the cohort study, prevalence and incidence of mental disorders (depression, anxiety, PTSD, somatisation and suicidality) will be assessed.
Phase 3: Odds ratios (with 95% confidence intervals) for factors associated with common mental disorders among perinatal and non-perinatal women | September 2023 - August 2024
  During the cohort study, risk factors associated with mental disorders (depression, anxiety, PTSD, somatisation and suicidality) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Gracia Fellmeth, DPhil, Principal Investigator — University of Oxford
Locations (2):
- India (2):
  - Dr Rajendra Prasad Government Medical College, Kangra, Himachal Pradesh
  - National Institute of Mental Health and Neuro Sciences, Bengaluru, Karnataka

IPD SHARING:
Plan to Share IPD: Undecided
Upon completion of the study, sharing of data with other researchers will be considered by the study team on a case-by-case basis. If data is shared this will not include any patient-identifying information.

REFERENCES:
- [Background] Fellmeth G, Kishore MT, Verma A, Desai G, Bharti O, Kanwar P, Singh S, Thippeswamy H, Chandra PS, Kurinczuk JJ, Nair M, Alderdice F. Perinatal mental health in India: protocol for a validation and cohort study. J Public Health (Oxf). 2021 Oct 8;43(Suppl 2):ii35-ii42. doi: 10.1093/pubmed/fdab162. PMID 34622290